CLINICAL TRIAL: NCT05039281
Title: Phase I/II Study to Evaluate the Safety and Clinical Efficacy of Atezolizumab (Anti-PD-L1) in Combination With Cabozantinib in Patients With Recurrent Glioblastoma (rGBM)
Brief Title: Atezolizumab and Cabozantinib for the Treatment of Recurrent Glioblastoma
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-0041; NCI-2021-09119 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2021-0041 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2021-09-01; First posted 2021-09-09 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Recurrent Glioblastoma; Recurrent Gliosarcoma
MeSH Terms: conditions — Glioblastoma; Gliosarcoma | interventions — atezolizumab; cabozantinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (atezolizumab, cabozantinib) (Experimental): Patients receive atezolizumab IV over 30-60 minutes on day 1 and cabozantinib PO on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Atezolizumab; Drug: Cabozantinib

INTERVENTIONS:
Biological: Atezolizumab — Given IV
  Other Names: MPDL 3280A; MPDL 328OA; MPDL-3280A; MPDL3280A; MPDL328OA; RG7446; RO5541267; Tecentriq
Drug: Cabozantinib — Given PO

SUMMARY:
This phase I/II trial tests the safety and side effects of atezolizumab in combination with cabozantinib and whether they work to shrink tumors in patients with glioblastoma that has come back (recurrent). Immunotherapy with monoclonal antibodies, such as atezolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Cabozantinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving atezolizumab and cabozantinib may help control the disease in patients with recurrent glioblastoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the safety of atezolizumab in combination with cabozantinib. (Phase I) II. To evaluate the progression-free survival at six months (PFS-6) of atezolizumab in combination with cabozantinib. (Phase II)

SECONDARY OBJECTIVE:

I. To evaluate the progression free survival (PFS), overall survival (OS), overall response rate (ORR) and duration of response of atezolizumab in combination with cabozantinib.

CORRELATIVE OBJECTIVES:

I. Profiling tumor immune cell populations (i.e., macrophage migration inhibitory factor [mIF] and immunohistochemistry [IHC] analyses of CD4, CD8, PD1, PD-L1, and PD-L2 expression).

II. Profiling of tumor, e.g., deoxyribonucleic acid (DNA), messenger (m) ribonucleic acid (RNA), microRNA and epigenetic profiling (DNA methylation), whole exome sequencing, RNA sequencing, and microRNA sequencing.

III. Peripheral blood collection for evaluation of circulating chemokines/cytokines.

IV. Stool collection for gut microbiome profiling.

OUTLINE:

Patients receive atezolizumab intravenously (IV) over 30-60 minutes on day 1 and cabozantinib orally (PO) once daily (QD) on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days, and then every 3 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent form (ICF)
* Ability and willingness to comply with the requirements of the study protocol
* Age >= 18 years
* Have histologically confirmed World Health Organization grade IV glioma (glioblastoma or gliosarcoma). Archival tissue will be required for diagnosis confirmation. Receipt of archival tissue is not required for the start of treatment
* Patients must have been previously treated with radiation and temozolomide
* Patients must be at least 12 weeks out from completion of concurrent chemoradiation
* Have a performance status of >= 60 on the Karnofsky performance status (KPS)
* Patients at either first or second recurrence will be considered eligible
* A baseline brain magnetic resonance imaging (MRI) obtained no more than 14 days prior to study enrollment
* Absolute neutrophil count (ANC) >= 1,500 /mcL
* Platelets >= 100,000 /mcL
* Hemoglobin >= 9 g/dL or >= 5.6 mmol/L
* Serum creatinine =< 1.5 X upper limit of normal (ULN) OR measured or calculated creatinine clearance (glomerular filtration rate [GFR] can also be used in place of creatinine or creatinine clearance [CrCl]) >= 60 mL/min for subject with creatinine levels > 1.5 X institutional ULN

  * Creatinine clearance should be calculated per institutional standard
* Urine protein/creatinine ratio (UPCR) =< 1 mg/mg (=< 113.2 mg/mmol) OR 24 hour (h) urine protein =< 1g
* Serum total bilirubin =< 1.5 X ULN OR direct bilirubin =< ULN for subjects with total bilirubin levels > 1.5 ULN
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamic pyruvic transaminase [SGPT]) =< 2.5 X ULN
* Serum albumin >= 2.8 g/dl
* International normalized ratio (INR) or prothrombin time (PT) activated partial thromboplastin time (aPTT) =< 1.3 X ULN
* All screening labs should be performed within 14 days (+3 working days) of treatment initiation
* Female subject of childbearing potential should have a negative serum pregnancy test within 14 days (+/- 3 working days) of study enrollment
* Female subjects of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the duration of the study and 5 months after the last dose of study treatment. Subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year
* Male subjects should agree to use an adequate method of contraception during the course of the study and 5 months after the last dose of study treatment

Exclusion Criteria:

* Has received prior interstitial brachytherapy, implanted chemotherapy, or therapeutics delivered by local injection or convection enhanced delivery. Prior treatment with Gliadel wafers will be excluded. Active treatment with the Optune device will be excluded
* Has received radiation therapy for bone metastasis within 2 weeks or any other radiation therapy within 4 weeks before first dose of study treatment, or systemic treatment with radionuclides within 6 weeks before first dose of study treatment
* Has clinically relevant ongoing complications from prior radiation therapy
* Is currently participating in any other recurrent therapeutic trial after completion of chemoradiation
* Has history of cavitating pulmonary lesion(s) or known endotracheal or endobronchial disease manifestation
* Any serious medical condition that interferes with adherence to study procedures
* Malignancies other than the disease under study within 5 years prior to cycle 1, day 1, with the exception of those with a negligible risk of metastasis or death and with expected curative outcome (such as adequately treated carcinoma in situ of the cervix, basal or squamous cell skin cancer, or ductal carcinoma in situ treated surgically with curative intent) or undergoing active surveillance per standard-of-care management (e.g., chronic lymphocytic leukemia Rai Stage 0)
* Has known leptomeningeal disease, gliomatosis cerebri, extracranial disease, or multifocal disease. Subject has multifocal glioblastoma (GBM), defined as discrete sites of contrast enhancing disease without contiguous T2/fluid attenuated inversion recovery (FLAIR) abnormality that require distinct radiotherapy ports. Satellite lesions that are associated with a contiguous area of T2/FLAIR abnormality as the main lesion(s) and that are encompassed within the same radiotherapy port as the main lesion(s) are permitted
* Has history of interstitial lung disease or active, non-infectious pneumonitis
* Has an active infection requiring systemic therapy
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the screening visit
* Contraindication for undergoing MRIs
* Inability to comply with study and follow-up procedures
* History or risk of autoimmune disease, including but not limited to systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Sjogren's syndrome, Bell's palsy, Guillain-Barre syndrome, multiple sclerosis, autoimmune thyroid disease, vasculitis, or glomerulonephritis

  * Patients with a history of autoimmune hypothyroidism on a stable dose of thyroid replacement hormone may be eligible
  * Patients with controlled type 1 diabetes mellitus on a stable insulin regimen may be eligible
  * Patients with eczema, psoriasis, lichen simplex chronicus of vitiligo with dermatologic manifestations only (e.g., patients with psoriatic arthritis would be excluded) are permitted provided that they meet the following conditions:

    * Patients with psoriasis must have a baseline ophthalmologic exam to rule out ocular manifestations
    * Rash must cover less than 10% of body surface area (BSA)
    * Disease is well controlled at baseline and only requiring low potency topical steroids (e.g., hydrocortisone 2.5%, hydrocortisone butyrate 0.1%, fluocinolone 0.01%, desonide 0.05%, aclometasone dipropionate 0.05%)
    * No acute exacerbations of underlying condition within the last 12 months (not requiring psoralen plus ultraviolet A radiation [PUVA], methotrexate, retinoids, biologic agents, oral calcineurin inhibitors; high potency or oral steroids)
* Has a medical history of idiopathic pulmonary fibrosis, pneumonitis (including drug induced), organizing pneumonia (i.e., bronchiolitis obliterans, cryptogenic organizing pneumonia, etc.), or active pneumonitis

  * History of radiation pneumonitis in the radiation field (fibrosis) is permitted
* Any other diseases, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that may affect the interpretation of the results or render the patient at high risk from treatment complications
* History of human immunodeficiency virus (HIV) infection or active hepatitis B (HBV) (chronic or acute) or hepatitis C infection

  * Patients with past or resolved hepatitis B infection (defined as having a negative hepatitis B surface antigen [HBsAg] test and a positive anti-HBc [antibody to hepatitis B core antigen] antibody test) are eligible. Patients will be sampled for HBV DNA and will be referred to a virologist to monitor for HBV re-activation
  * Patients positive for hepatitis C virus (HCV) antibody are eligible only if polymerase chain reaction (PCR) is negative for HCV RNA
* Active tuberculosis
* Severe infections within 4 weeks prior to cycle 1, day 1, including but not limited to hospitalization for complications of infection, bacteremia, or severe pneumonia
* Signs or symptoms of infection within 2 weeks prior to cycle 1, day 1
* Received oral or IV antibiotics within 2 weeks prior to cycle 1, day 1

  * Patients receiving prophylactic antibiotics (e.g., for prevention of a urinary tract infection or chronic obstructive pulmonary disease) are eligible
* Anticipation of need for a major surgical procedure (e.g., laparoscopic nephrectomy, gastrointestinal [GI] surgery, removal or biopsy of brain metastasis) within 2 weeks before first dose of study treatment, or of need for a minor surgery within 10 days before first dose of study treatment. Subjects must have complete wound healing from major surgery or minor surgery before first dose of study treatment. Subjects with clinically relevant ongoing complications from prior surgery are not eligible
* Administration of a live, attenuated vaccine within 4 weeks before cycle 1, day 1 or anticipation that such a live, attenuated vaccine will be required during the study
* Influenza vaccination should be given during influenza season only (approximately October to March). Patients must not receive live, attenuated influenza vaccine (e.g., FluMist) within 4 weeks prior to cycle 1, day 1 or at any time during the study and for 5 months after last dose of atezolizumab
* Patients may not receive concomitant chemotherapy, hormonal therapy, immunotherapy, or radiotherapy while patients are on study
* MEDICATION-RELATED EXCLUSION CRITERIA:
* Prior treatment with anti-PD-1, or anti-PD-L1 therapeutic antibody or pathway-targeting agents
* Receipt of any type of cytotoxic, biologic or other systemic anticancer therapy (including investigational) within 4 weeks before first dose of study treatment
* Receipt of any type of small molecule kinase inhibitor (including investigational kinase inhibitor) within 2 weeks before first dose of study treatment
* Prior treatment with anti-angiogenic (e.g. anti-vascular endothelial growth factor [VEGF]) therapeutic antibody or pathway targeting agents
* Treatment with systemic immunostimulatory agents (including but not limited to interferon [IFN]- or interleukin [IL]-2) within 6 weeks or five half-lives of the drug (whichever is shorter) prior to cycle 1, day 1
* Treatment with systemic immunosuppressive medications (including but not limited to prednisone, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor [anti-TNF] agents) within 2 weeks prior to cycle 1, day 1

  * Patients who have received acute, low-dose, systemic immunosuppressant medications (e.g., a one-time dose of dexamethasone for nausea) may be enrolled
  * The use of inhaled corticosteroids and mineralocorticoids (e.g., fludrocortisone) for patients with orthostatic hypotension or adrenocortical insufficiency is allowed
* History of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies, fusion proteins or components of cabozantinib
* Patients with prior allogeneic bone marrow transplantation or prior solid organ transplantation
* Evidence of recent hemorrhage on post-operative MRI of the brain, however patients with clinically asymptomatic presence of hemosiderin, resolving post-operative changes and punctate intratumoral hemorrhage are permitted
* Known lesions invading or encasing any major blood vessels. Subjects with lesions invading the intrahepatic vasculature, including portal vein, hepatic vein, and hepatic artery, are eligible
* Corrected QT interval calculated by the Fridericia formula (QTcF) > 500 ms per electrocardiogram (ECG) within 14 days before first dose of study treatment

  * Note: if a single ECG shows a QTcF with an absolute value > 500 ms, two additional ECGs at intervals of approximately 3 min must be performed within 30 minutes after the initial ECG, and the average of these three consecutive results for QTcF will be used to determine eligibility
* Inability to swallow tablets
* Inadequately controlled hypertension (defined as systolic blood pressure > 140mmHg and/or diastolic blood pressure > 90mmHg)
* A history of or active nephrotic syndrome
* Prior history of hypertensive crisis or hypertensive encephalopathy
* New York Heart Assocation (NYHA) grade II or greater congestive heart failure
* History of myocardial infarction or unstable angina within 6 months prior to study enrollment
* History of stroke or transient ischemic attack (TIA) within 6 months prior to study enrollment
* Significant vascular disease (e.g. aortic aneurysm requiring surgical repair or recent peripheral arterial thrombosis) within 6 months prior to study enrollment
* History of clinically significant hematuria, hematemesis, or hemoptysis of > 0.5 teaspoon (2.5 ml) of red blood, or any other history of significant bleeding (e.g. pulmonary hemorrhage) within 12 weeks before first dose of study treatment
* Evidence of bleeding diathesis or coagulopathy (in the absence of therapeutic anticoagulation)
* Major surgical procedure, open biopsy, intracranial biopsy, ventriculoperitoneal shunt or significant traumatic injury within 28 days prior to study enrollment
* Core biopsy (excluding intracranial biopsy) or other minor surgical procedure within 107 days prior to study enrollment. Placement of a central vascular access device if performed within 2 days prior to cabozantinib administration
* History of abdominal fistula, bowel obstruction, gastrointestinal perforation or intra-abdominal abscess within 6 months before first dose of study treatment

  * Note: complete healing of an intra-abdominal abscess must be confirmed before first dose of study treatment
* History of tumor invading the GI tract, active peptic ulcer disease, inflammatory bowel disease (e.g., Crohn's disease), diverticulitis, cholecystitis, symptomatic cholangitis or appendicitis, acute pancreatitis, acute obstruction of the pancreatic duct or common bile duct, or gastric outlet obstruction
* History of intracranial abscess within 6 months prior to study enrollment
* Clinically-significant disorders that would preclude safe study participation

  * Serious non-healing wound, active ulcer or untreated bone fracture
  * Uncompensated/symptomatic hypothyroidism
  * Moderate to severe hepatic impairment (Child-Pugh B or C)
* Concomitant anticoagulation with coumarin agents (e.g., warfarin), direct thrombin inhibitors (e.g. , dabigatran), direct factor Xa inhibitor betrixaban, or platelet inhibitors (e.g., clopidogrel)

  * Prophylactic use of low-dose aspirin for cardio-protection (per local applicable guidelines) and low-dose low molecular weight heparins (LMWH) are allowed
  * Therapeutic doses of LMWH or anticoagulation with direct factor Xa inhibitors rivaroxaban, edoxaban, or apixaban in subjects without known brain metastases who are on a stable dose of the anticoagulant for at least 1 week before first dose of study treatment without clinically significant hemorrhagic complications from the anticoagulation regimen or the tumor are also allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2022-09-23 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | At 6 momths
  Will estimate the 6 months PFS distribution using the Kaplan-Meier method.
Objective response rate | Up to 3 years
  Will be estimated with exact binomial 95% confidence intervals. Logistic regression will be used to explore the correlations between response rates and correlative markers.
Incidence of adverse events | Up to 3 years
  Will be estimated with exact binomial 95% confidence intervals. Adverse events will be tabulated by grade and by their relationship to the treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Shiao-Pei S Weathers, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org